CLINICAL TRIAL: NCT01973868
Title: A Phase 1b, Multi-center, Non-randomized, Open Label, Dose Escalation Design Study of Regorafenib (BAY73-4506) in Combination With Cetuximab in Subjects With Locally Advanced or Metastatic Solid Tumors Who Are Not Candidates for Standard Therapy or in Whom Regorafenib or Cetuximab is Considered as a Standard Treatment
Brief Title: Safety and Pharmacokinetics of Regorafenib and Cetuximab in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16547
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms
Keywords: Regorafenib; Cetuximab; Solid tumors; Cancer; Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — regorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib will be administered once daily on Days 1-21 of each 28-day Cycle (3 weeks on / 1 week off). The starting dose of regorafenib is 120 mg q.d., if this is tolerable in combination with cetuximab the dose will be escalated to 160 mg q.d.; if it is not tolerated the dose will be de-escalated to 80 mg q.d.
  Subjects will receive an initial i.v. infusion of cetuximab (loading dose of 400 mg/ m2 BSA) on Pre-cycle Day -7.
  The treatment of regorafenib in combination with cetuximab maintenance dose (250 mg/m2 BSA) starts on Cycle 1 Day 1.
  Cetuximab infusions will be given in a once-weekly dosing-regimen as approved.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Cetuximab (ERBITUX)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506)
Drug: Cetuximab (ERBITUX)

SUMMARY:
To establish safety, tolerability and pharmacokinetics of regorafenib and cetuximab in combination, and to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed, locally advanced or metastatic solid tumors who are not candidates for standard therapy or in whom regorafenib or cetuximab is considered a standard treatment. Patients with metastatic colorectal cancer (mCRC) must have a record of K-ras gene mutational analysis available and no K-ras mutation is present.
* Male or female patients ≥ 18 years of age
* Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements conducted within 7 days of starting the study treatment:

  * Platelet count ≥ 100,000/cubic millimeters (mm3), hemoglobin (Hb) ≥ 8.5 g/dl, leukocyte count > 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,000/mm3
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN). Mildly elevated total bilirubin (< 6 mg/dL) is allowed if Gilbert's syndrome is documented.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects whose cancer involves their liver).
  * Amylase and lipase ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 times ULN and creatinine clearance (CLcr) ≥ 30 mL/min according to the Cockroft-Gault formula
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Prior treatment with Regorafenib
* Prior discontinuation of cetuximab treatment due to toxicity or intolerance of cetuximab
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
* Non-healing wound, ulcer, or bone fracture
* Systemic anticancer therapy within 28 days
* Patients unable to swallow and retain oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of regorafenib in combination with cetuximab | 1 month
  MTD is defined as the maximum dose at which the incidence of dose-limiting toxicities (DLTs) during Cycle 1 is below 20 %, or as the maximum dose administered, whichever is achieved first during dose escalation
Number of participants with Adverse Events as a measure of safety and tolerability | Up to 2 years or longer
Cmax,md (Cmax after multiple dose) for regorafenib and cetuximab | Multiple time points on Day 15
AUC(0-24)md (AUC from time zero to 24 hours after multiple-dose administration) for regorafenib | Multiple time points on Day 15
AUC(0-26)md (AUC from time zero to 26 hours after multiple-dose administration) for cetuximab | Multiple time points on Day 15

SECONDARY OUTCOMES:
Tumor response according to RECIST 1.1 | Up to 2 years or longer
tmax,md (tmax after multiple-dose administration) for regorafenib, its metabolites M-2 (BAY75-7495) and M-5 (BAY81-8752) and cetuximab | Multiple time points on Day 15
tlast,md (tlast after multiple dosing) for regorafenib, its metabolites M-2 (BAY75-7495) and M-5 (BAY81-8752) and cetuximab | Multiple time points on Day 15
Cmax,md for metabolites M-2 (BAY75-7495) and M-5 (BAY81-8752) | Multiple time points on Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Weekes C, Lockhart AC, Lee JJ, Sturm I, Cleton A, Huang F, Lenz HJ. A phase 1b study evaluating the safety and pharmacokinetics of regorafenib in combination with cetuximab in patients with advanced solid tumors. Int J Cancer. 2019 Nov 1;145(9):2450-2458. doi: 10.1002/ijc.32317. Epub 2019 Jun 14. PMID 30958892